# Statistical analysis plan

# Nurse-led Smoking Cessation Intervention with Follow-up in Healthy Life Centers: a Randomized Clinical Trial

# **Table of content**

| 1. | Administrative information | 3 |
|---|---|---|
| | 1.1 Trial registration numbers | 3 |
| | 1.2 Protocol version used for preparation of the statistical analysis plan | 3 |
| | 1.3 Contributors for preparation of the statistical analysis plan | 3 |
| | 1.4 Signatures | 3 |
| | 1.5 SAP Revision | 3 |
| 2. | Introduction | 4 |
| | 2.1 Background and rationale for the study | 4 |
| | 2.2 Objectives | 5 |
| | 2.2.1 Primary objective | 5 |
| | 2.2.2 Secondary objectives | 5 |
| | 2.2.3 Exploratory objectives | 5 |
| | 2.2.4 Secondary and exploratory objectives for future sub-studies | 6 |
| 3. | Study methods | 6 |
| | 3.1 Trial design and randomization | 6 |
| | 3.2 Intervention | 6 |
| | 3.3 Framework, sample size and power calculation | 6 |
| | 3.4 Interim analysis for effect | 7 |
| | 3.5 Timing of final analysis and outcome assessments | 7 |
| 4. | Statistical principles | 7 |
| | 4.1 Confidence interval and P values | 7 |
| | 4.2 Protocol deviations | 7 |
| | 4.3 Analysis population | 7 |
| 5. | Trial population | 7 |
| | 5.1 Screening | 7 |
| | 5.2 Inclusion and exclusion criteria | 8 |
| | 5.3 Information to be included in the CONSORT flow diagram | 8 |
| | 5.4 Withdrawal and loss to follow-up | 8 |
| | 5.4.1 Withdrawal of informed content | 8 |
| | 5.4.2 Loss to follow up | 8 |

| | 5.5 Data collection | 8 |
|---|---|---|
| | 5.6 Patient characteristics in main publication | 9 |
| 6. | Analysis and endpoints | 10 |
| | 6.1 Endpoints | 10 |
| | 6.1.1 Primary endpoint | 10 |
| | 6.1.2 Secondary endpoints | 10 |
| | 6.1.3 Exploratory endpoints | 10 |
| | 6.1.4 Secondary and exploratory endpoints for future sub-studies | 11 |
| | 6.2 Analyses | 11 |
| | 6.2.1 Analysis of the primary endpoint | 11 |
| | 6.2.2 Analyses of key secondary endpoints | 11 |
| | 6.2.3 Additional analyses | 11 |
| | 6.2.4 Planned subgroup analyses | 11 |
| | 6.2.5 Secondary and exploratory endpoints and data to be included in sub studies | 12 |
| | 6.3 Missing data | 13 |
| | 6.4 Harms | 13 |
| | 6.4.1 Safety endpoints | 13 |
| | 6.4.2 Adverse events | 13 |
| | 6.4.3 Details of guidelines for stopping the trial early | 13 |
| 7. | Data handling and record keeping | 13 |
| 8. | Supplementary materials | 14 |
| | Study protocol evaluated by the ethics committee (ref. number: 270267) and the Data protection officer (ref. number: 21/07103-1 / 005) version 2.0, 31.08. 21 (in Norwegian) | 14 |
| 9. | | |

#### 1. Administrative information

The "Nurse-led Smoking Cessation Intervention with Follow-up in Healthy Life Centers: a Randomized Clinical Trial" aims to investigate clinical and health economic effects of a multi-component intervention for smoking cessation following an atherosclerotic cardiovascular disease event.

# 1.1 Trial registration numbers

This is a (ClinicalTrials.gov Identifier: NCT05049174) multicenter trial that enroll patients from three hospitals within the Vestre Viken Health Trust.

# 1.2 Protocol version used for preparation of the statistical analysis plan Protocol version 2.0, 24.08.2022.

#### 1.3 Contributors for preparation of the statistical analysis plan

Project leader/main supervisor John Munkhaugen and PhD candidate Karin Pleym Statisticians: Harald Weedon-Fekjær and Morten Wang Fagerland (QC)

The SAP has been approved by the NORCOR smoking cessation project steering committee including user representatives.

# 1.4 Signatures

| Project leader | PhD student |
|----------------------------|-----------------------------|
| Name: John Munkhaugen | Name: Karin Pleym |
| Signature: | Signature: |
| Date: | Date: |
| Study Statistician | QC statistician |
| Name: Harald Weedon-Fekjær | Name: Morten Wang Fagerland |
| Signature: | Signature: |
| Date: | Date: |

# 1.5 SAP Revision

| Date of revision | Revision | Justification for revision |
|---|---|---|
| 06.03.2024 | Health-economic analysis in a separate paper | After careful discussions with leading national healtheconomists, we agreed that a comprehensive Markow analysis needs to be elaborated in a separate paper and not included in the main publication. |

#### 2. Introduction

# 2.1 Background and rationale for the study

Cigarette smoking is a major risk factor for numerous diseases including atherosclerotic cardiovascular disease (ASCVD).<sup>1-3</sup> The detrimental health effects from smoking lead to extended disability and premature mortality, quantifiable by disability-adjusted life-years (DALYs).<sup>4</sup> In 2019, tobacco smoking was responsible for more than 7 million deaths and 200 million DALYs worldwide.<sup>5</sup> These figures underscore the substantial burden tobacco smoking places on individuals, healthcare systems, and society at large.<sup>6,7</sup>

Smoking cessation following an ASCVD event mitigates the likelihood of subsequent vascular events and mortality. However, cessation rates remain modest or low among patients with various presentations of ASCVD. However, cessation rates remain modest or low among patients with various presentations of ASCVD. However, cessation rates remain modest or low among patients with a stroke or those smoking preceding an unplanned coronary heart disease event continued smoking after hospital discharge. Correspondingly, up to 60% of smoking patients hospitalized with a stroke or transient ischemic attack (TIA) continue to smoke. A recent study revealed that more than 70% of patients with peripheral artery disease were daily smokers one year after hospitalization. Of these, only 1 in 5 were referred to formal cessation counseling and 1 in 10 were prescribed smoking cessation drugs. Thus, it is crucial to establish and implement smoking cessation interventions across vascular diagnoses. Extensive evidence for the effectiveness of pharmacological and behavioural smoking cessation measures is available. However, implementing this knowledge into clinical practice remains challenging due to individual and systemic barriers.

The majority of smoking ASCVD patients have a long history of smoking and come from socio-economically disadvantaged backgrounds. <sup>20-22</sup> Low socio-economic status is associated with low health literacy which in turn may pose a significant barrier to seeking, finding and participating in relevant smoking cessation programs. <sup>23,24</sup> Notably, more than 70% of daily smokers express a desire to quit. <sup>25</sup> An acute ASCVD event and subsequent hospitalization may act as a catalyst for these patients, enhancing their motivation for smoking cessation. <sup>26</sup> In this setting, healthcare providers have an unique opportunity to identify smokers and provide tailored counselling and support. <sup>27</sup> Importantly, smoking cessation interventions for hospitalized patients should extend for a minimum of one month after discharge. <sup>28</sup> This knowledge encourages care coordination between specialist and primary health care.

Unfortunately, only a small minority of ASCVD patients in Norway and Europe currently access or participate in cardiac rehabilitation programs.<sup>29,30</sup> Within the Norwegian primary healthcare system, community-based Healthy Life Centers take part in preventive care alongside general practitioners and cardiac rehabilitation services.<sup>31,32</sup> These centers offer a variety of health-promoting measures, including smoking cessation programs providing cessation drugs at no cost.<sup>33</sup> Patients can initiate contact with the Healthy Life Center themselves, but also be referred by healthcare professionals for participation.

Based on key factors known to promote successful smoking cessation,<sup>34-37</sup> we developed a nurse-led, multi-component cessation intervention tailored for smokers hospitalized with acute ASCVD events. The intervention builds on existing infrastructure of the Norwegian healthcare system. The purpose was to enhance cessation rates by capitalizing on the possible increased readiness to quit

related to hospitalization.<sup>26</sup> Accordingly, the intervention began during hospital stay with nurse-led cessation counseling, employing recommended motivational interviewing techniques.<sup>34,38</sup> Furthermore, we aimed to provide a seamless transition to post-discharge follow-up care in community-based Healthy Life Center smoking cessation programs.<sup>35</sup> Thus, nurses actively referred patients by telephone to their local community-based center for continued follow-up. Moreover, staff members from Healthy Life Centers proactively contacted the patient by telephone, inviting them to participate in the cessation program. We hypothesized that this strategy would effectively promote smoking cessation among patients hospitalized with ASCVD. We anticipated that the impact of the intervention would be mediated through motivational counseling, proactive referral, increased participation in smoking cessation programs, and increased use of cessation drugs.

In a recent feasibility study, we assessed the effect of this intervention on participation rate and use of cessation drugs.<sup>39</sup> Compared to the control group, the nurse-led intervention significantly increased participation in the Healthy Life Center cessation programs, with a 48% participation rate versus 7% in the control group. Additionally, the use of cessation drugs was significantly higher in the intervention group.<sup>39</sup> An exploratory evaluation showed promising results in smoking cessation at six months, with 48% of the intervention group successfully quitting compared to 25% in the control group.<sup>39</sup> Despite the small sample size (N=58), these encouraging results call for a larger-scale, statistically robust trial to determine the effectiveness of the intervention. The primary objective of this pragmatic randomized study is to determine the effect of the multi-component nurse-led intervention on smoking cessation rates at six- and 12 months follow-up after an ASCVD event. Additionally, we aim to conduct a cost-effectiveness analysis of the intervention.

#### 2.2 Objectives

The overall aim is to evaluate the clinical and health economic effects of a nurse-led, multi-component intervention tailored to daily smokers admitted to the hospital with an acute ASCVD event.

#### 2.2.1 Primary objective

To determine the effect of the multi-component nurse-led intervention on self-reported smoking cessation rates at six-month follow-up.

# 2.2.2 Secondary objectives

# **Key secondary objective:**

To determine the effect of the intervention on smoking cessation verified by carbon monoxide measurements in exhaled breathing air at six-month follow-up.

#### Other Secondary objectives:

- **#1.** To determine differences between the groups in participation rate at the cessation program.
- **#2.** To determine differences in self-reported use of cessation drugs between the groups.
- **#3.** To determine the effect of the intervention on smoking cessation at 12 months follow-up.

# 2.2.3 Exploratory objectives

- **#1.** To determine differences in self-reported smoking cessation rates at six-month follow-up in the following subgroups; age, sex, ASCVD diagnosis, somatic comorbidity, and study site.
- **#2.** To explore between-group differences in the composite end-point of all-cause mortality and unplanned re-hospitalizations for ASCVD events (i.e. myocardial infarction, angina/claudication, coronary and peripheral revascularization procedures, stroke/TIA, tachyarrhythmia's and/or heart failure).

# 2.2.4 Secondary and exploratory objectives for sub-studies

The following objectives pertain to sub-studies planned for subsequent publications.

- **#1.** To perform a cost-effectiveness analysis of the intervention.
- **2.** To explore between-group differences in the composite end-point of all-cause mortality and unplanned re-hospitalizations for ASCVD events at 5- and 10-years follow-up.
- **#3.** Investigate whether baseline levels and longitudinal changes in the following PROMs are associated with smoking cessation between treatment arms and in the entire study cohort:
  - Symptoms of depression, anxiety, insomnia, and sleep duration.
  - Type D personality.
  - Metacognitions (as measured by DTQ, MSQ, MCQ-30).
- **#4.** Identify clinical and psychosocial predictors of smoking cessation in a combined analysis, incorporating data from the current trial (N=220) and the pilot study (N=58).

#### 3. Study methods

#### 3.1 Trial design and randomization

This is a prospective, randomized, multi-center, parallel-group, open-label, blinded end-point (PROBE) clinical trial evaluating the effect of a multi-component smoking cessation intervention. Patients will be randomized 1:1 to the multi-component intervention or to usual care plus an information leaflet. The randomization will be stratified by study site. The three study sites are Drammen hospital, Kongeberg hospital and Ringerike hospital.

#### 3.2 Intervention

The multi-component intervention includes 1) counselling utilizing motivational interview technique, 2) an information-leaflet, 3) referral to a post-discharge municipal smoking cessation program providing access to free nicotine replacement therapy, 4) a proactive invitation by telephone to participation in the cessation program after hospital discharge and 5) a letter to the general practitioner informing about the inclusion in the study and the option of participating in the Healthy Life center for smoking cessation. The control group received treatment and follow-up care according to routine clinical practice at the participating hospitals and in primary care plus an information-leaflet describing the cessation program and how to initiate contact for participation.

#### 3.3 Framework, sample size and power calculation

The trial will be analyzed as an ordinary superiority trial and is designed to have more than 90% power to detect a between-group difference of 23% (48% vs. 25%) in occurrence of the primary outcome, self-report smoking cessation at six months follow-up (with an alpha of 0.05). The difference is based on results for our pilot study conducted in 2021 (ClinicalTrials.gov Identifier:

NCT04772144). With 196 (98 x2) patients we also have 80% power to detect an even more conservative difference in point prevalence of smoking cessation of 19% (44% vs. 25%) between treatment groups. To account for slightly lower effects of the intervention, we will randomize 220 patients. The database will be locked and the study un-blinded when the last randomized patients have been followed for a minimum of 6 months.

# 3.4 Interim analysis for effect

No interim analyses are planned.

# 3.5 Timing of final analysis and outcome assessments

The final analyses will be performed when follow-up has ended, and all endpoints have been registered and after database lock. The minimum follow-up period will be 6 months.

Primary, secondary and exploratory endpoints are collected from 1) medical records at the participating hospitals and community-based cessation centers at study end, 2) telephone interviews conducted after one, three, six- and 12-months follow-up, 3) self-report questionnaires collected at baseline and at six months after randomization, and 4) carbon monoxide (CO) measurements collected six months after randomization.

# 4. Statistical principles

#### 4.1 Confidence intervals and P values

For the primary outcome we will use a significance level of 5% and a confidence interval (CI) of 95% will be reported. The secondary outcomes will be assessed with a CI of 95%. All statistical tests and confidence intervals will be two-sided.

#### 4.2 Protocol deviations

Possible protocol deviations are linked to situations where:

- The patient refuse to participate in the motivational interview conversation
- The nurse for some reason do not refer the patient to community-based Healthy Life
- The Healthy Life Center fail to pro-actively contact the patient and inviting them to participate

Should such situations occur, they will be registered.

### 4.3 Analysis population

All major comparisons between the randomized groups will be performed according to the principle "intention-to-treat", i.e., participants will be analyzed, and endpoints counted in the group to which they were assigned at randomization.

#### 5. Trial population

# 5.1 Screening

Patients admitted to the hospital for an ASCVD event will be screened for inclusion and exclusion criteria at all participating centers. All sites in are consecutively reporting the reasons for not being included in the trial. Collected screening data will be summarized and presented in the main publication.

#### Screening data registered in the eCRF of all screened patients:

- Site
- Exclusion criteria (see below)

#### 5.2 Inclusion and exclusion criteria

| Inclusion criteria | • >18 years |
|---|---|
| | Smoking at least one cigarette daily |
| | <ul> <li>Hospitalized with an acute cardiovascular disease event and established<br/>atherosclerosis (based on diagnosis and/or treatment with a lipid<br/>lowering and antiplatelet)</li> </ul> |
| <b>Exclusion criteria</b> | Patients not living in or working in the Vestre Viken region |
| | Any condition (psychosis, alcohol abuse, dementia) or situation that may pose a significant risk to the participant, or make participation unethical |
| | Short life expectancy (<12 months) |
| | Not able to understand and write Norwegian |
| | Decline to participate |

#### 5.3 Information to be included in the CONSORT flow diagram

- Number of patients assessed for eligibility
- Number of patients excluded and reason for exclusion
- Number of patients randomized
- Number of patients allocated to the intervention or the control group
- Number of loss to follow-up
- Number of patients excluded from analyses and reasons for exclusion

# 5.4 Withdrawal and loss to follow-up

#### 5.4.1 Withdrawal of informed content

Patient consent withdrawals are possible at any time during follow-up and the day of withdrawal will be registered. Time to withdrawal will be summarized.

#### 5.4.2 Loss to follow up

All non-responders will be categorized as current smokers in the primary analysis according to the Russel criteria.<sup>40</sup>

#### 5.5 Data collection

#### Data collected from hospital medical records at baseline:

- Demographics
- Information about the qualifying ASCVD event treatment and/or procedures performed during index event
- Major comorbidities summarized into Charlson comorbidity score
- Risk factors

# Patient reported outcomes measures collected at baseline and after six months follow-up:

**a. Socio-economic variables:** Education, employment status, marital status (living alone or with others)

- **b. Smoking history and behavior:** cigarettes/day, number of years daily smoking, previous quit attempts, smoking partner, motivation to quit (readiness for smoking cessation), nicotine addiction (Fagerstrøm), previous use of nicotine replacement therapy and/or ecigarettes.
- c. Lifestyle: Physical activity, alcohol consumption, height and weight calculated into BMI
- **d. Other post-discharge follow-up**: participation in cardiac rehabilitation, follow-up with GP.
- e. Screening question for quality of life: SF-12- Question 1.
- **f. Measures of depression and anxiety**: HADS (Hospital Anxiety and Depression Scale)
- g. Measures of sleeping disorder: Bergen insomnia Scale and average sleep duration
- h. Measures of personality: Type D (distressed) personality disorder.
- i. Measures of metacognitions: Desired Thinking Questionnaire (DTQ; Spada & Caselli, 2011), Metacognitions about smoking questionnaire (MSQ; Nikcevic, Caselli, Wells & Spada, 2015) and Metacognition Questionnaire-30 (MCQ-30)

#### Data collected during follow-up:

Primary, secondary and safety endpoints are collected through questionnaires, medical records at participating hospitals and municipality centers, CO measurements, and telephone interviews throughout the trial as previously described.

#### 5.6 Patient characteristics in main publication

#### Data at baseline:

- Demographics and social background
  - Age, sex, marital status/living condition (living alone, living with partner or in a care home facility), employment status and education level
- Index cardiovascular event
  - Acute myocardial infarction/stroke vs. other atherosclerotic cardiovascular disease events
- Somatic comorbidities, risk factors and treatment
  - Hypertension (diagnosis and/or treatment), hyperlipidemia (treatment with statins and/or ezetimibe), chronic kidney disease, diabetes (diagnosis/treatment), physical inactivity, alcohol consumption, obesity, antiplatelet
  - Previous cardiovascular disease, Charlson comorbidity score
  - HADS-Score
- Quality of life -single screening questionSmoking frequency, history and motivation
  - Nicotine dependency
    - Fagerstrøms test
    - Time to first cigarette
  - Duration of smoking
  - Living with a daily smoker
  - Previous quit attempt and eventually use of nicotine replacement therapy and/or ecigarettes.

- Motivation to quit on a 0-10 Likert scale
- Readiness for smoking cessation
  - Preparation phase, contemplation phase, pre-contemplation phase

#### Follow-up care after discharge

- Participation in cardiac rehabilitation
- Visits to general practitioner
- Participation in Healthy Life Center

#### Details of how baseline characteristics will be descriptively summarized

Baseline characteristics will be presented as numbers with percentages for categorical variables and medians with interquartile ranges for continuous variables.

#### 6. Analysis and endpoints

# 6.1 Endpoints

# 6.1.1 Primary endpoint

Difference between the groups in the proportion of participants who self-report smoking abstinence at six months follow-up.

#### 6.1.2 Secondary endpoints

#### *Key secondary endpoint:*

Difference between the groups in the proportion of participants who self-report smoking abstinence at six months follow-up verified by carbon monoxide (CO) measurements in the exhaled air, according to the Russel standard.<sup>40</sup>

#### Other secondary endpoints:

- **#1.** The proportion of participants who self-report smoking abstinence at 12 months follow-up.
- **#2.** Participation rate at the cessation program between the groups obtained from medical records at the municipal centers at six months follow-up.
  - Number of consultations per participant (digital vs. physical)
  - Number of individual and group-based consultations per participant
  - O Number of vouchers (for 4 weeks use of cessation drugs) delivered (0 to 3) per participant
- **#3.** Patient report use of cessation drugs between the groups at six months follow-up.

# 6.1.3 Exploratory endpoints

The following exploratory endpoint will be included in the main publication:

- **#1.** The proportion of participants who self-report smoking abstinence at six months follow-up in clinical subgroups as specified in 6.2.4.
- **#2.** Time to all-cause mortality or myocardial infarction, unplanned re-hospitalizations for cardiovascular disease events (i.e. angina/claudication, revascularization procedures, stroke/TIA, arrhythmia and/or heart failure) obtained from hospital medical records after three and five years follow-up.

# 6.1.4 Secondary and exploratory endpoints for future sub-studies

Planned analyses of other secondary and exploratory endpoints for future sub studies are described under 6.2.5.

# 6.2 Analyses

# 6.2.1 Analysis of the primary endpoint

The primary assessment will use an intention-to-treat approach among all randomized participants to evaluate the effects of group allocation on the primary endpoint. Main secondary analyses will use an intention-to-treat approach to evaluate the effects of intervention allocation on the proportion of secondary endpoints among all randomized participants.

The primary endpoint is the proportion who self-report smoking cessation assessed after the last patient included has completed 6 months of follow-up. The null hypothesis is that the proportion of the primary endpoint in the allocation groups are equal. The primary analysis will be a binary logistic regression model with randomization group as the main covariate. The analysis will be adjusted for site (the stratification factor in the randomization). An odds ratio (OR) for intervention vs control group with a 95% confidence interval (CI) will be estimated, and a P-value for the null hypothesis of a odds ratio equal to 1 will be computed.

#### Decision rule:

- If the estimated OR is > 1 and the 95% CI does not contain 1, superiority of the intervention will be accepted.
- If the estimated OR is < 1 and the 95% CI does not contain 1, superiority of the control group will be accepted.
- If the 95% CI contains 1, no superiority will be accepted

#### 6.2.2 Analyses of secondary endpoints

The key secondary endpoint and other secondary endpoints to be included in the main publication are listed in section 6.1.2. All dichotomous end-points will be analyzed in the same manner as the primary endpoint, except only the CI will be computed and reported, and not the P-value. Secondary discrete numerical endpoints (mean number of events per participant) will be analyzed with linear regression models, where randomized group and site will be covariates. The estimated difference (intervention - control) with a 95% CI will be reported. The health economic analysis are detailed in 6.2.3.

#### 6.2.3 Additional analyses

Exploratory analysis: Numeric differences in (first and all) recurrent cardiovascular events and all-cause mortality between the intervention and control group will be summarized. Due to an expected high probability of type II error, no statistical comparisons are planned.

#### 6.2.4 Planned subgroup analyses

The following subgroup analyses of the primary study end point are planned in the primary publication:

- Age (</≥ median age)</li>
- Gender (male vs. female)
- Charlson comorbidity score (</≥ median score)</li>
- Acute myocardial infarction or stroke vs. other ASCVD events

- Study site (Drammen vs. Kongsberg vs. Ringerike)

The subgroup analyses will be performed by adding an interaction term in the logistic regression model (as described in Section 6.2.1) between the intervention and the subgroup-defining factor. A P-value ≤ 0.05 for the interaction term will indicate a significant subgroup effect. An OR with 95% CI for intervention vs. control group will be estimated for each subgroup and presented in a forest plot. For age and Charlson comorbidity score, the lowest category will be reference value.

<u>Exploratory analyses in the main publication</u>: Nicotine dependency (Fagerstøm score), Readiness for cessation (Stages of change), motivation (0-10 Likert scale), smoking partner, HADS-score Anxiety and Depression.

#### 6.2.5 Secondary and exploratory endpoints and data to be included in sub studies

The following data will be used in sub studies planned for later publications. Study data and planned analyses are not elaborated in detail as these will not be included in the main publication.

# #1 Health economic cost-effectiveness analysis:

We will assess the cost-effectiveness of the intervention using a Markov model. Health outcomes will be recurrent ASCVD events, COPD, pneumonia, and quality-adjusted life years (QALYs). Costs and health-outcomes will be assessed in a lifetime-perspective for the treatment and control group. To establish the effectiveness of our intervention, we will consider the proportion of patients who self-report smoking abstinence in both groups. The latest available data from our study will inform these proportions.

At the 6-month evaluation point, we will rely on existing literature to establish our outcome rates, because the 6-month timeframe may be insufficient for accurately assessing the risk of recurrent ASCVD events. At the 22 months, 5- and 10-year cutoff points, we will incorporate data from our ongoing study. At 22 months follow-up, we will compare estimates from the observed study data and the literature to evaluate if follow up time is sufficient.

Unit costs related to outcomes will be based on diagnosis-related groups (DRGs) and their weights. 41 QALYs will be informed by the existing literature and monetized following national guidelines. 42

The primary cost associated with our nurse-led intervention is the time spent counseling patients in the treatment group. We will calculate the unit cost of the intervention by considering the wages for nurses, including associated social costs, and the time invested in counseling and patient follow-up.

In a supplementary analysis we will assess the cost-effectiveness of free cessation drugs.

Our analysis will include the calculation of an incremental cost-effectiveness ratio (ICER) compared to multiple predefined thresholds, in alignment with established guidelines.

- **#2.** Time to all-cause mortality or unplanned re-hospitalizations for cardiovascular disease events obtained from hospital medical records at 5- and 10-years follow-up.
- **#3.** Differences between the groups in the proportion of participants who self-report smoking abstinence at six- and 12 months follow-up.

# 6.3 Missing data

Follow-up is through medical records, telephone interviews, and self-report questionnaires as previously described. We anticipate no missing data on the primary or main secondary outcomes since non-responders to the six-month follow-up interview will be classified as smokers according to the Russel standard.<sup>40</sup> We therefore do not plan to replace missing data in the main publication.

#### 6.4 Harms

# 6.4.1 Safety endpoints

The primary components of the intervention which is motivational interviewing and a pro-active referral approach do not have effects that could cause any harm to participants. However all patients will have access to free nicotine replacement therapy (NRT) if they choose to participate in the community-based smoking cessation offer. The main concern with NRT in ASCVD patients is that nicotine can elevate heart rate and blood pressure. However, the levels of nicotine provided by NRT are usually lower and more stable than the spikes from inhaling cigarette smoke. Furthermore, clinical guidelines indicates that NRT can be used safely in patients with cardiovascular disease who are trying to quit smoking. Thus, no safety analyses are planned.

#### 6.4.2 Adverse events

All unplanned hospitalizations and all-cause death, including potential endpoints, will be registered from hospital medical records

Tables summarizing adverse events:

- All-Cause Mortality:
- Total number of hospitalizations
- Descriptive statistics will be displayed for continuous data and for categorical data.

# 6.4.3 Details of guidelines for stopping the trial early

The steering committee recommended not to set any criteria for early termination of the trial as all participants has equal access to the community-based smoking cessation program regardless of group assignment.

# 7. Data handling and record keeping

Data is collected for participants who enter the randomized phase of the study. All source data will be entered into an electronic data system (Ledidi). The dataset will be prepared and stored at the secured research server in Vestre Viken Trust. This dataset forms the basis for all statistical analyses, which will be performed by the study statisticians in collaboration with the QC statistician. The Oslo Center for Biostatistics and Epidemiology will perform internal database quality-control checks.

# 8. Supplementary materials

Study protocol evaluated by the ethics committee (ref. number: 270267) and the Data protection officer (ref. number: 21/07103-1 / 005) version 2.0, 31.08. 21 (in Norwegian).

#### 9. References

- 1. Dai X, Gakidou E, Lopez AD. Evolution of the global smoking epidemic over the past half century: strengthening the evidence base for policy action. *Tob Control* 2022;**31**:129-137. doi: 10.1136/tobaccocontrol-2021-056535
- 2. Visseren FLJ, Mach F, Smulders YM, et al. 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice. *Eur Heart J* 2021;**42**:3227-3337. doi: 10.1093/eurheartj/ehab484
- 3. Arnett DK, Blumenthal RS, Albert MA, et al. 2019 ACC/AHA guideline on the primary prevention of cardiovascular disease: a report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. *Circulation* 2019;**140**:e596-e646. doi:
- 4. Reitsma MB, Kendrick PJ, Ababneh E, *et al.* Spatial, temporal, and demographic patterns in prevalence of smoking tobacco use and attributable disease burden in 204 countries and territories, 1990–2019: a systematic analysis from the Global Burden of Disease Study 2019. *The Lancet* 2021;**397**:2337-2360. doi: DOI:https://doi.org/10.1016/S0140-6736(21)01169-7
- 5. Goodchild M, Nargis N, Tursan d'Espaignet E. Global economic cost of smoking-attributable diseases. *Tob Control* 2018;**27**:58-64. doi: 10.1136/tobaccocontrol-2016-053305
- 6. Steen Carlsson K, Nilsson K, Wolden ML, Faurby M. Economic burden of atherosclerotic cardiovascular disease: a matched case-control study in more than 450,000 Swedish individuals. *BMC Cardiovasc Disord* 2023;**23**:483. doi: 10.1186/s12872-023-03518-y
- 7. Ekpu VU, Brown AK. The Economic Impact of Smoking and of Reducing Smoking Prevalence: Review of Evidence. *Tob Use Insights* 2015;**8**:1-35. doi: 10.4137/tui.S15628
- 8. Ding N, Sang Y, Chen J, et al. Cigarette Smoking, Smoking Cessation, and Long-Term Risk of 3 Major Atherosclerotic Diseases. *J Am Coll Cardiol* 2019;**74**:498-507. doi: 10.1016/j.jacc.2019.05.049
- 9. Kotseva K, Wood D, De Backer G, et al. Cardiovascular prevention guidelines in daily practice: a comparison of EUROASPIRE I, II, and III surveys in eight European countries. *The Lancet* 2009;**373**:929-940. doi:
- 10. Wechsler PM, Liberman AL, Restifo D, *et al.* Cost-Effectiveness of Smoking Cessation Interventions in Patients With Ischemic Stroke and Transient Ischemic Attack. *Stroke* 2023;**54**:992-1000. doi: doi:10.1161/STROKEAHA.122.040356
- 11. Patel KK, Jones PG, Ellerbeck EF, et al. Underutilization of evidence-based smoking cessation support strategies despite high smoking addiction burden in peripheral artery disease specialty care: insights from the international PORTRAIT registry. *Journal of the American Heart Association* 2018;**7**:e010076. doi:
- 12. De Bacquer D, Astin F, Kotseva K, et al. Poor adherence to lifestyle recommendations in patients with coronary heart disease: results from the EUROASPIRE surveys. European Journal of Preventive Cardiology 2021;**29**:383-395. doi: 10.1093/eurjpc/zwab115
- 13. Patel KK, Jones PG, Ellerbeck EF, et al. Underutilization of Evidence-Based Smoking Cessation Support Strategies Despite High Smoking Addiction Burden in Peripheral Artery Disease Specialty Care: Insights from the International PORTRAIT Registry. *Journal of the American Heart Association* 2018;**7**:e010076. doi: 10.1161/jaha.118.010076
- 14. Hartmann-Boyce J, Ordóñez-Mena JM, Livingstone-Banks J, *et al.* Behavioural programmes for cigarette smoking cessation: investigating interactions between behavioural, motivational and delivery components in a systematic review and component network meta-analysis. *Addiction* 2022;**117**:2145-2156. doi: https://doi.org/10.1111/add.15791
- 15. Rice VH, Heath L, Livingstone-Banks J, Hartmann-Boyce J. Nursing interventions for smoking cessation. *Cochrane Database Syst Rev* 2017;**12**:Cd001188. doi: 10.1002/14651858.CD001188.pub5

- 16. Stead LF, Koilpillai P, Fanshawe TR, Lancaster T. Combined pharmacotherapy and behavioural interventions for smoking cessation. *Cochrane Database of Systematic Reviews* 2016. doi: 10.1002/14651858.CD008286.pub3
- 17. Andrew LP, William E, Sophia P. Smoking cessation: health system challenges and opportunities. *Tobacco Control* 2022;**31**:340. doi: 10.1136/tobaccocontrol-2021-056575
- 18. Getz V, Munkhaugen J, Lie HC, Dammen T. Barriers and facilitators for smoking cessation in chronic smokers with atherosclerotic cardiovascular disease enrolled in a randomized intervention trial: A qualitative study. *Frontiers in Psychology* 2023;**14**. doi: 10.3389/fpsyg.2023.1060701
- 19. Nielsen JB, Leppin A, Gyrd-Hansen DE, *et al.* Barriers to lifestyle changes for prevention of cardiovascular disease a survey among 40-60-year old Danes. *BMC Cardiovasc Disord* 2017;**17**:245. doi: 10.1186/s12872-017-0677-0
- 20. Sverre E, Otterstad JE, Gjertsen E, et al. Medical and sociodemographic factors predict persistent smoking after coronary events. *BMC Cardiovascular Disorders* 2017;**17**:241. doi: 10.1186/s12872-017-0676-1
- 21. Ohm J, Kuja-Halkola R, Warnqvist A, et al. Socioeconomic Disparities and Mediators for Recurrent Atherosclerotic Cardiovascular Disease Events After a First Myocardial Infarction. *Circulation* 2023;**148**:256-267. doi: 10.1161/circulationaha.123.064440
- 22. Gregoraci G, Lenthe FJv, Artnik B, *et al.* Contribution of smoking to socioeconomic inequalities in mortality: a study of 14 European countries, 1990–2004. *Tobacco Control* 2017;**26**:260-268. doi: 10.1136/tobaccocontrol-2015-052766
- 23. Brørs G, Dalen H, Allore H, et al. Health Literacy and Risk Factors for Coronary Artery Disease (From the CONCARD(PCI) Study). *Am J Cardiol* 2022;**179**:22-30. doi: 10.1016/j.amjcard.2022.06.016
- 24. Svendsen MT, Bak CK, Sørensen K, et al. Associations of health literacy with socioeconomic position, health risk behavior, and health status: a large national population-based survey among Danish adults. *BMC Public Health* 2020;**20**:565. doi: 10.1186/s12889-020-08498-8
- 25. Joly B, Perriot J, d'Athis P, et al. Success rates in smoking cessation: Psychological preparation plays a critical role and interacts with other factors such as psychoactive substances. *PLoS One* 2017;**12**:e0184800. doi: 10.1371/journal.pone.0184800
- 26. Riley H, Ainani N, Turk A, *et al.* Smoking cessation after hospitalization for myocardial infarction or cardiac surgery: Assessing patient interest, confidence, and physician prescribing practices. *Clin Cardiol* 2019;**42**:1189-1194. doi: 10.1002/clc.23272
- 27. Sharpe T, Alsahlanee A, Ward KD, Doyle F. Systematic Review of Clinician-Reported Barriers to Provision of Smoking Cessation Interventions in Hospital Inpatient Settings. *Journal of Smoking Cessation* 2018;**13**:233-243. doi: 10.1017/jsc.2017.25
- 28. Rigotti NA, Clair C, Munafò MR, Stead LF. Interventions for smoking cessation in hospitalised patients. *Cochrane Database Syst Rev* 2012;**5**:Cd001837. doi: 10.1002/14651858.CD001837.pub3
- 29. Norekvål TM, Bale M, Bedane HK, *et al.* Cardiac rehabilitation participation within 6 months of discharge in 37 136 myocardial infarction survivors: a nationwide registry study. *European Journal of Preventive Cardiology* 2023. doi: 10.1093/eurjpc/zwad350
- 30. Ruivo J, Moholdt T, Abreu A. Overview of Cardiac Rehabilitation following post-acute myocardial infarction in European Society of Cardiology member countries. *Eur J Prev Cardiol* 2023;**30**:758-768. doi: 10.1093/eurjpc/zwad024
- 31. Helsedirektoratet. Healthy Life Centres in Norway <a href="https://www.helsedirektoratet.no/english/healthy-life-centres">https://www.helsedirektoratet.no/english/healthy-life-centres</a> (25.03.2022 2022)
- 32. Peersen K, Munkhaugen J, Gullestad L, *et al.* The role of cardiac rehabilitation in secondary prevention after coronary events. *European Journal of Preventive Cardiology* 2017;**24**:1360-1368. doi: 10.1177/2047487317719355
- 33. Helsedirektoratet. Tobakksfri. Mal for snus- og røykesluttkurs for deg som jobber på frisklivsetralen. In; 2012, 48.

- 34. Lindson N, Thompson TP, Ferrey A, Lambert JD, Aveyard P. Motivational interviewing for smoking cessation. *Cochrane Database of Systematic Reviews* 2019. doi: 10.1002/14651858.CD006936.pub4
- 35. van Westen-Lagerweij NA, Hipple Walters BJ, Potyka F, Croes EA, Willemsen MC. Proactive referral to behavioral smoking cessation programs by healthcare staff: a systematic review. *Nicotine & Tobacco Research* 2022. doi:
- 36. Hartmann-Boyce J, Chepkin SC, Ye W, Bullen C, Lancaster T. Nicotine replacement therapy versus control for smoking cessation. *Cochrane Database of Systematic Reviews* 2018. doi: 10.1002/14651858.CD000146.pub5
- 37. Vibjerg H. The Danish model for smoking cessation. *Tobacco Prevention & Cessation* 2021;**7**. doi: 10.18332/tpc/143631
- 38. Rollnick S, Miller WR, Butler C. Motivational interviewing in health care: helping patients change behavior. Second edition ed: The Guilford Press; 2022.
- 39. Pleym K, Sverre E, Weedon-Fekjaer H, et al. Effect of in-hospital nurse-led smoking cessation intervention for patients with atherosclerotic cardiovascular disease: a randomised pilot study. European Heart Journal 2022;**43**. doi: 10.1093/eurheartj/ehac544.2329
- 40. West R, Hajek P, Stead L, Stapleton J. Outcome criteria in smoking cessation trials: proposal for a common standard. *Addiction* 2005;**100**:299-303. doi: 10.1111/j.1360-0443.2004.00995.x
- 41. Helsedirektoratet. DRG-systemet. https://www.helsedirektoratet.no/tema/finansiering/innsatsstyrt-finansiering-og-drg-systemet/drg-systemet (29.09.2023 2023)
- 42. Legemiddelverk. S. Guidelines for the submission of documentation for single technology assessment (STA) of pharmaceuticals.

https://legemiddelverket.no/Documents/English/Public%20funding%20and%20pricing/Documentation%20for%20STA/Guidelines%2018.10.2021.pdf (29.09.2023 2023)